CLINICAL TRIAL: NCT02259374
Title: Use of Tap Block in Patients After Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Principal Investigator, thong sze ying, ASSOCIATE CONSULTANT, Singapore General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014/729/D
Record Dates: First submitted 2014-09-30; First posted 2014-10-08 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Abdominal Hysterectomy (& Wertheim)
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAP BLOCK 0.2% ROPIVACAINE (Active Comparator): Patients randomised into this group will receive bilateral TAP block (single shot) with 0.2% ropivacaine after hysterectomy.
  Intervention: TAP block Dose: 20 ml 0.2% ropivacaine
  Interventions: Procedure: TAP BLOCK 0.2% ROPIVACAINE; Procedure: TAP BLOCK 0.4% ROPIVACAINE
- TAP BLOCK 0.4% ROPIVACAINE (Active Comparator): Patients randomised into this group will receive bilateral TAP block (single shot) with 0.4% ropivacaine after hysterectomy.
  Intervention: TAP block Dose: 20 ml 0.4% ropivacaine
  Interventions: Procedure: TAP BLOCK 0.2% ROPIVACAINE; Procedure: TAP BLOCK 0.4% ROPIVACAINE

INTERVENTIONS:
Procedure: TAP BLOCK 0.2% ROPIVACAINE — Patients randomised to this group will receive 20 ml 0.2% Ropivacaine for bilateral TAP block after hysterectomy
Procedure: TAP BLOCK 0.4% ROPIVACAINE — Patients randomised to this group will receive 20 ml 0.4% Ropivacaine for bilateral TAP block after hysterectomy

SUMMARY:
TAP block performed under ultrasound guidance is used as part of multimodal analgesia to relieve pain after abdominal surgery in our hospital. Choices of local anaesthetic used include bupivacaine and ropivacaine. Local anaesthetic works by inhibiting nerve transmission of pain from the site of tissue injury. An important component of the pain experienced by patients after abdominal surgery derives from the abdominal wall incision. The abdominal wall sensory afferents course through the transversus abdominis (neurofascial) plane superficial to the transversus abdominis muscle. Single shot TAP block has been shown to provide pain relief of up to 24h in surgeries involving pfannenstiel incisions, hence a study period of 24h is chosen in patients undergoing hysterectomy.

This study was designed to test the hypothesis that the TAP block, as part of a multimodal analgesic regimen, even at a lower concentration, would provide effective analgesia in the first 24 h after hysterectomy, in comparison to a higher concentration of 0.4% ropivacaine.

DETAILED DESCRIPTION:
Our study hypothesis is that TAP block performed with 0.2% ropivacaine is not inferior to that using 0.4% ropivacaine.

The primary outcome measure in this study was 24 h morphine consumption. Secondary outcome measures included time to first request for morphine, VAS scores, and side effects associated with morphine consumption which include nausea, vomiting, sedation, pruritus, as well as patient satisfaction.

Our study hypothesis is that TAP block performed with 0.2% ropivacaine 40ml is not inferior to that using 0.4% ropivacaine 40ml, in terms of analgesia in the first 24h.

Primary Objectives Morphine consumption in the first 24h should not differ between the 2 groups by more than 10mg.

Secondary Objectives Secondary objectives are to show that morphine side effects are similar in the two groups if a lower ropivacaine provides similar pain relief as higher concentration. Patient satisfaction is also recorded.

54 patients undergoing hysterectomy will be recruited from SGH.

Criteria for Recruitment and Recruitment Process Patients will be shortlisted from the surgical list the week prior to surgery. Patients seen in the pre anaesthetic assessment clinic will also be invited to take part in the study. A simple history and physical assessment will determine eligibility. Patients fitting the inclusion criteria will be approached for the study with the emphasis that participation is voluntary and refusal to participate will not affect subsequent conduct of anaesthesia or care. Patient's wishes will be respected should she request not to participate

STUDY DESIGN Double blind randomise control trial. Study design is non-inferiority trial testing 0.2% ropivacaine vs 0.4% ropivacaine. Expected 1 year to complete recruitment of 54 patients. All patients are expected to participate in the study for a period of 24h and will be followup during their convalescence in the hospital. There will be no change in scheduling of operation or additional visits for the purpose of the study.

Ultrasound images of the block may be stored in the thumb drive. However, the images will not be linked to patient identifiers. It will be stored in password protected thumb drive and kept in the department under lock and key.

It may be used for illustration if the research is published in a scientific journal.

Randomisation and Blinding Patients will be randomised into of the 2 groups - 0.2% or 0.4% ropivacaine group. The allocation sequence will be generated by a random number table, and group allocation will be concealed in sealed, opaque envelopes, which will not be opened until just prior to block performance.

The anaesthesiologist performing the block and anaesthesia will not be blinded. However, the patient, surgeon and researcher collecting subsequent patient data will be blinded.

Randomisation code will be broken after the final analysis of the study results. As both study groups involve the use of ropivacaine at concentration below the maximum recommended dose, the likelihood of needing to break the randomisation code is low. However, should that become necessary, the study PI can break the code.

Study Visits and Procedures Study visit 1: recruitment during pre-anaesthesia visit a day before surgery Procedure: Bilateral TAP block after surgery, before reversal of anaesthesia. Followup for 24h, which includes 1 study visit to elicit pain scores and side effects of opioids.

Screening Visits and Procedures History and physical examination are required to evaluate recruitment criteria. Patients will be invited to participate in the study after meeting inclusion criteria.

Study Visits and Procedures

1 visit in the post operative period.

Final Study Visit:

Patient will be seen once after operation in the first post operative day to assess for VAS scores, and side effects associated with morphine consumption which include nausea, vomiting, sedation, pruritus, as well as patient satisfaction.

Post Study Follow up and Procedures Patient will be seen once after operation in the first post operative day to assess for VAS scores, and side effects associated with morphine consumption which include nausea, vomiting, sedation, pruritus, as well as patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* - ASA 1-3
* age 21-60
* undergoing open hysterectomy as planned by the surgeons
* able to provide informed consent. A upper limit age of 60 is chosen because elderly patients may have reduced requirements for analgesia and may be more sensitive to effects of opioids.

Exclusion Criteria:

* - chronic pain/ opioid usage
* allergy to study drugs
* BMI>35
* Weight <50

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption in the first 24 hours | 24hours

SECONDARY OUTCOMES:
Morphine side effects | 24 hours
Patient satisfaction | 24 hours